CLINICAL TRIAL: NCT02497196
Title: Neurophysiological Effects on tPCS and tDCS on Healthy Subjects and on Patients With Chronic Visceral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Prinicipal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015P000365
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Visceral Pain; Pancreatitis; Pelvic Pain
Keywords: TPCS; tDCS; visceral pain; pancreatitis; healthy subjects; pelvic pain; neuromodulation; non-invasive brain stimulation
MeSH Terms: conditions — Visceral Pain; Pancreatitis; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part 1:Active tPCS, Active tDCS (Experimental): 12 out of the 48 total health subjects will receive active tPCS and active tDCS. This will be done for 20 minutes simultaneously.
  Interventions: Device: Active tPCS; Device: Active tDCS
- Part 1: Active tPCS, Sham tDCS (Experimental): 12 out of the 48 total health subjects will receive active tPCS and sham tDCS. This will be done for 20 minutes simultaneously.
  Interventions: Device: Active tPCS; Device: Sham tDCS
- Part 1:Sham tPCS, Active tDCS (Experimental): 12 out of the 48 total health subjects will receive sham tPCS and active tDCS. This will be done for 20 minutes simultaneously.
  Interventions: Device: Active tDCS; Device: Sham tPCS
- Part 1: Sham tDCS, Sham tDCS (Sham Comparator): 12 out of the 48 total health subjects will receive sham tPCS and sham tDCS. This will be done for 20 minutes simultaneously.
  Interventions: Device: Sham tPCS; Device: Sham tDCS
- Part 2: Active tPCS/Active tDCS (Experimental): Part 2 will run as a four-period crossover design, where all chronic visceral pain subjects (18 total) will be receiving all (4) possible combinations of tDCS and tPCS interventions (active or sham) at the end of the experiment in a random, consecutive way. This represents the combination of receiving active tPCS and active tDCS (1/4 combinations all subjects will receive).
  Interventions: Device: Active tPCS; Device: Active tDCS
- Part 2: Active tPCS/Sham tDCS (Experimental): Part 2 will run as a four-period crossover design, where all chronic visceral pain subjects (18 total) will be receiving all (4) possible combinations of tDCS and tPCS interventions (active or sham) at the end of the experiment in a random, consecutive way. This represents the combination of receiving active tPCS and sham tDCS (1/4 combinations all subjects will receive).
  Interventions: Device: Active tPCS; Device: Sham tDCS
- Part 2: Sham tPCS/Active tDCS (Experimental): Part 2 will run as a four-period crossover design, where all chronic visceral pain subjects (18 total) will be receiving all (4) possible combinations of tDCS and tPCS interventions (active or sham) at the end of the experiment in a random, consecutive way. This represents the combination of receiving sham tPCS and active tDCS (1/4 combinations all subjects will receive).
  Interventions: Device: Active tDCS; Device: Sham tPCS
- 2: Sham tPCS/Sham tDCS (Sham Comparator): Part 2 will run as a four-period crossover design, where all chronic visceral pain subjects (18 total) will be receiving all (4) possible combinations of tDCS and tPCS interventions (active or sham) at the end of the experiment in a random, consecutive way. This represents the combination of receiving sham tPCS and sham tDCS (1/4 combinations all subjects will receive).
  Interventions: Device: Sham tPCS; Device: Sham tDCS

INTERVENTIONS:
Device: Active tPCS — A current intensity of 2mA and a stimulation frequency range of 6-10 Hz will be used with a peri-aurical ear-clip electrode montage for 20 minutes.
  Arms: Part 1: Active tPCS, Sham tDCS; Part 1:Active tPCS, Active tDCS; Part 2: Active tPCS/Active tDCS; Part 2: Active tPCS/Sham tDCS
Device: Active tDCS — A current intensity of 2.0 mA will be used for 20 minutes. The electrodes that will be used will be standard sponge electrodes. The anode will be placed over left motor cortex. The cathode electrode will be placed over the contralateral supraorbitofrontal area.
  Arms: Part 1:Active tPCS, Active tDCS; Part 1:Sham tPCS, Active tDCS; Part 2: Active tPCS/Active tDCS; Part 2: Sham tPCS/Active tDCS
Device: Sham tPCS — Sham tPCS stimulation will consist of applying the same parameters as for active, but the corresponding device will be turned off after 30 seconds, as to simulate the initial sensation of the active current. A current intensity of 2mA and a stimulation frequency range of 6-10 Hz will still be used (only this will be turned off after 30 seconds using ramping) with a peri-aurical ear-clip electrode montage.
  Arms: 2: Sham tPCS/Sham tDCS; Part 1: Sham tDCS, Sham tDCS; Part 1:Sham tPCS, Active tDCS; Part 2: Sham tPCS/Active tDCS
Device: Sham tDCS — Sham tDCS stimulation will consist of applying the same parameters as for active, but the corresponding device will be turned off after 30 seconds, as to simulate the initial sensation of the active current. A current intensity of 2.0 mA will still be used (but turned off after 30 seconds using ramping). The electrodes that will be used will be same, standard sponge electrodes. The anode will be placed over the left motor cortex The cathode electrode will be placed over the contralateral supraorbitofrontal area.
  Arms: 2: Sham tPCS/Sham tDCS; Part 1: Active tPCS, Sham tDCS; Part 1: Sham tDCS, Sham tDCS; Part 2: Active tPCS/Sham tDCS

SUMMARY:
This study investigates comparing the effects of transcranial Pulsed Current Stimulation and transcranial Direct Current Stimulation (tDCS) (Soterix ©) and their combination on neurophysiological outcomes on healthy subjects as well as on the clinical population for chronic visceral pain. The study also aims to evaluate the effects of these techniques on pain thresholds in healthy subjects as well as for chronic visceral pain patients.

ELIGIBILITY:
PART 1: 48 healthy subjects will be selected to take part in this study. All healthy subjects will need to meet all of the following inclusion criteria and none of the following exclusion criteria:

Inclusion criteria:

* Provide informed consent to participate in the study
* Age 18 - 60 years

Exclusion criteria:

* History of alcohol or substance abuse within the last 6 months as self-reported
* Severe depression (with a score of >30 in the Beck Depression Inventory)*
* History of seizures during the last two years or diagnosis of epilepsy
* History of neurological or psychiatric illness
* Unstable medical conditions such as uncontrolled diabetes mellitus, uncompensated cardiac pathology, heart failure, kidney insufficiency or chronic obstructive pulmonary disease, acute thrombosis
* History of head injury resulting in more than a momentary loss of consciousness during the last two years
* History of unexplained fainting spells or loss of consciousness as self-reported during the last two years
* Contraindication to tPCS or tDCS
* Metallic brain implants
* Implanted brain electronic medical devices
* Pregnancy
* Use of neuropsychotropic drugs within the past two weeks as self reported

Part 2: 18 patients with Chronic Visceral Pain will take part in this experiment. All subjects must meet the following criteria:

Inclusion criteria:

* Provide informed consent to participate in the study
* Age 18 - 60 years
* Abdominal or pelvic pain for ≥ 3 days per week for at least 3 months (average VAS scale score of 4/10 or greater at time of enrollment) as self reported
* Diagnosis of chronic visceral pain (e.g. Chronic Pancreatitis or Chronic Pelvic Pain) as confirmed by medical records or a letter from their physician
* If taking pain medications, stable doses are required for at two weeks prior to initiation of the study

Exclusion criteria:

* History of alcohol or substance abuse within the last 6 months as self-reported
* Severe depression (with a score of >30 in the Beck Depression Inventory)*
* Epilepsy
* Unstable medical conditions such as uncontrolled diabetes mellitus, uncompensated cardiac pathology, heart failure, kidney insufficiency or chronic obstructive pulmonary disease, acute thrombosis
* History of head injury resulting in more than a momentary loss of consciousness during the last two years
* History of unexplained fainting spells or loss of consciousness as self-reported during the last two years
* Contraindication to tPCS or tDCS
* Metallic brain implants
* Implanted brain electronic medical devices
* Pregnancy or trying to become pregnant during the next month
* Use of carbamazepine oxcarbazepine, phenytoin, pramipexole (Mirapex), or cavergoline (Dostinex) within the past 6 months as self-reported

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-07; Primary Completion 2016-10-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Signal Coherence and EEG power as measured Quantitative Electroencephalographic Analysis (qEEG): | For the healthy subjects during their 1-time study visit; For visceral pain patients, it will be measured over the course of about 3 weeks
  The EEG test is performed to measure the electrical activity in the brain and to examine the dynamic changes.

SECONDARY OUTCOMES:
Pressure Values as measured by Pain Pressure Test (PPT) for Conditioned Pain Modulation (CPM) | For the healthy subjects during their 1-time study visit; For visceral pain subjects, it will be measured over the course of about 3 weeks
  These procedures incorporate a conditioning stimulus (a noxious stimulus that evokes Descending Noxious Inhibitory Control (DNIC) activation) and a test stimulus (a noxious stimulus used to evaluate the analgesic response to the conditioning stimulus- this will be the PPT as determined by an algometer (JTECH medical)). This study will evaluate CPM in healthy subjects as well as in patients with chronic visceral pain using pressure as the test stimulus, and cold water as the conditioning stimulus.
Sensitivity of Filaments as measured by Von Frey assessment | Only done for visceral pain subjects; it will be measured over the course of about 3 weeks.
  This assessment will be performed before and after every intervention on a patient with pain. Mechanical perception and pain threshold will be tested on the painful region and on other non-painful area Von Frey monofilaments (0.4 g to 50 g) (these are fine filaments that can test a subject's perception threshold when they are applied to the body surface). Monofilament application will be applied to the painful region and a non painful region on the same side of the body (i. e. left or right). The hairs will be applied until subject perceives the stimulus (perception threshold) and describes it as painful (pain threshold). The threshold will be taken as the lowest force that causes pain perception in the affected and contralateral mirror healthy site.
Pain score as measured by Visual Analogue Scale (VAS) for Pain: | Only done for visceral pain subjects; it will be measured over the course of about 3 weeks.
  The VAS is a self-reporting test asking subjects to self-measure their pain on a visual scale from zero to ten (i.e., none to unbearable). This will help us monitor changes in subjects' pain levels when they come in for sessions.
Pain levels and medication intake as measured Pain/Medication Diary | Only done for visceral pain subjects; it will be measured over the course of about 3 weeks
  To monitor pain levels, as well as safety, patients with chronic visceral pain will keep a diary listing their daily medications and pain levels when not at the laboratory.
Mood scores as measured Visual Analog Mood Scale (VAMS) | Only done for visceral pain subjects; it will be measured over the course of about 3 weeks
  This is a self-reporting assessment in which subjects rate their own emotions, including anxiety, depression, stress, and sleepiness along a 100mm line.
Depression level as measured Beck Depression Inventory (BDI) | Done for both healthy and visceral pain subjects during screening (first study visit)
  A 21-item, multiple-choice questionnaire will be administered at the beginning of the study to all subjects to assess the presence and degree of depression in adults, as studies in chronic pain have found that depression can modulate pain perception.
Effectiveness of blinding as measured by the tPCS and tDCS Blinding Questionnaire | For the healthy subjects during their 1-time study visit; For visceral pain subjects, it will be measured over the course of about 3 weeks
  After the stimulation session, subjects will complete a questionnaire to determine if the blinding methods were effective. A 30s sham montage is used,which is consistent with other trials, keeping the device on the subject for the duration of the session.
Side-effects from stimulation as measured by the tDCS and tPCS Side Effects Questionnaire | For the healthy subjects during their 1-time study visit; For visceral pain subjects, it will be measured over the course of about 3 weeks
  At the end of each stimulation session, subjects will complete a questionnaire to evaluate potential side effects of stimulation (headache, neck pain, mood alterations, and seizures) on a 5-point scale. Subjects will be asked whether they have experienced any side effects in open-ended questions. They will also be specifically asked about headache, neck pain, scalp pain, scalp burns, tingling, skin redness, sleepiness, trouble concentrating, and acute mood change. If any side effects are reported, the degree of relatedness to the intervention will be assessed.This assessment identifies adverse effects using open-ended questions.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, MPH, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Network Research Institute, Charlestown, Massachusetts, United States